CLINICAL TRIAL: NCT06541184
Title: Ziconotide for Non-cancer Pain by Intrathecal Administration
Status: Recruiting | Type: Observational
Sponsor: ESTEVE Pharmaceuticals SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: ZENITH
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pain, Chronic
Keywords: ziconotide; intrathecal analgesia; non-cancer pain; severe chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — ziconotide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated by ziconotide-based intrathecal analgesia (ITA): Patients followed during 2 years after an initiation of ziconotide. These patients will be recruited retrospectively or prospectively.
  Interventions: Drug: Ziconotide [Prialt]

INTERVENTIONS:
Drug: Ziconotide [Prialt] — Intrathecal injection of ziconotide, using an internal pump, surgically inserted by a trained neurosurgeon or anesthesiologist, under general anesthesia.

SUMMARY:
Although ziconotide's marketing authorization does not restrict its use to a given type of pain, the drug has been used mainly in cancer patients. Most data on ziconotide-based intrathecal (IT) treatment has therefore been obtained in this population, for whom the drug's place is clearly documented (national and international recommendations).

In contrast the management of non-cancer pain is less straightforward, partly because of the very large range of possible clinical conditions, and the utilization of ziconotide is poorly documented, mainly described in single-centre small series.

Due to the lack of data, physicians are often reluctant to undertake this type of treatment, which may represent a loss of opportunity for patients.

This registry aims at providing information on patients suffering from non-cancer pain refractory to standard therapy, treated by ziconotide-based intrathecal analgesia.

Patients suffering from all types of non-malignant pain will be eligible for the study, including but not limited to spinal cord injury, radiculopathy, failed back surgery, diabetic neuropathy, central pain syndrome, complex regional pain syndrome, chemotherapy-induced neuropathy, fibromyalgia.

The collected data will cover the first 2 years of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years,
2. Chronic non-cancer pain requiring interventional techniques, and eligible to ziconotide-containing intrathecal therapy,
3. Having received information on and not opposed to data collection,

Inclusion criteria specific for the retrospective cohort:

Currently treated by ziconotide-based ITA according to SmPC whatever the duration of treatment

Inclusion criteria specific for the prospective cohort:

Naïve of ITA and candidate to ziconotide-based ITA or already treated by IT route without ziconotide, scheduled for addition of ziconotide in the pump

Exclusion Criteria:

1. Contraindication to intrathecal therapy or to ziconotide
2. Any condition that may jeopardize appropriate follow-up of the treatment
3. Patient under guardianship or deprived of liberty by a judicial or administrative decision or unable to express opposition to data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic non-cancer pain requiring interventional techniques, and eligible to ziconotide-containing intrathecal therapy.
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2029-10-30 (Estimated); Study Completion 2029-10-30 (Estimated)

PRIMARY OUTCOMES:
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: demographic characteristics | Baseline (treatment initiation)
  Patient's demographic characteristics
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: medical history | Baseline (treatment initiation)
  Relevant medical history, including history of psychiatric disorders
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: indication for intrathecal ziconotide | Baseline (treatment initiation)
  Indication for ziconotide initiation (mechanism of pain and etiology)
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: starting date of pain | Baseline (treatment initiation)
  Starting date of severe/disabling pain
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: history of pain management | Baseline (treatment initiation)
  History of pain management including prior interventional techniques and current analgesic treatment (administered when decision of ziconotide treatment is made)
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: pain intensity | Baseline (treatment initiation)
  Numerical Rating Scale score for pain (graduated from 0: absence of pain to 10: worst possible pain) analgesic treatment (administered when decision of ziconotide treatment is made)
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: neuro-psychiatric condition | Baseline (treatment initiation)
  NPI-ES score (NeuroPsychiatric Inventory of An inventory of 12 of the most frequent symptoms of Alzheimer's disease and related disorders, assessing their frequency and severity, as well as the impact on the caregiver or professional), or score of another type or neuropsychological evaluation questionnaire)
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: disability condition | Baseline (treatment initiation)
  Owestry disability index score: patient-completed questionnaire which gives a subjective percentage score of level of function (disability) in 10 activities of daily living
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: anxiety and depression disorders | Baseline (treatment initiation)
  Hospital Anxiety and Depression Scale (HADS) score: patient-completed questionnaire with 14 items assessing anxiety and depressive disorders
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: reasons for initiating ziconotide | Baseline (treatment initiation)
  Reasons for initiating ziconotide (process of medical decision)
Describe the characteristics of patients treated by intrathecal ziconotide for chronic non-cancer pain: planned modification of the current intrathecal treatment | Baseline (treatment initiation)
  Planned modification of the current intrathecal treatment

SECONDARY OUTCOMES:
Describe the modalities of ziconotide therapy at ziconotide initiation | Baseline (treatment initiation)
  Ziconotide initial dose, concentration in the pump, administration in monotherapy or in combination, planned titration schedule, and concomitant non-IT analgesics.
Describe the modalities of ziconotide therapy during follow-up | 2 years follow-up
  Drugs added in or removed from the mixture ; Ziconotide posology and concentration in the pump, or ziconotide discontinuation; Evaluation of dose efficacy; Concomitant non-IT analgesics
Describe the patient's care pathway and treatment management | 2 years follow-up
  Characteristics of the physician who includes the patient; Decision to administer ziconotide in multidisciplinary meeting (MDM) and MDM members if applicable or specialty of the physician who made the decision if no MDM was organized; Type of investigations performed at inclusion and/or during follow-up (NPI-ES score or other type of neuropsychiatric evaluation), Owestry disability index, Hospital Anxiety and Depression Scale; Data on pump implantation
Describe the effect of treatment on pain evolution | 2 years follow-up
  Numerical Rating Scale (NRS) score graduated from 0 (absence of pain) to 10 (worst possible pain) collected at each visit, from inclusion to last visit
Describe the effect of treatment on disability | 3 months, 1 year and 2 years.
  Owestry disability index
Describe the effect of treatment on anxiety and depression | 3 months, 1 year and 2 years.
  Hospital Anxiety and Depression Scale score
Describe the safety and tolerability of treatment | From treatment initiation to 2 years of follow-up
  Adverse events, related to the intrathecal administration procedure or to the ziconotide

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Clinique de la Casamance, Aubagne
  - Hospices Civils de Lyon, Bron
  - Polyclinique du Parc, Caen
  - CHD Vendée, La Roche-sur-Yon
  - CH Laon, Laon
  - CHU Lille, Lille
  - Clinique Mutualiste de la Porte de l'Orient, Lorient
  - Centre Léon Bérard, Lyon
  - Hopital Saint Joseph, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CH Yves Le foll, Saint-Brieuc
  - CHU St Etienne, Saint-Etienne
  - IUCT Toulouse, Toulouse